CLINICAL TRIAL: NCT03605108
Title: The Influence of Oral Probiotics on the Microbiome and Lipidome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1242039
Record Dates: First submitted 2018-07-03; First posted 2018-07-30 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Gut Microbiome; Skin Microbiome; Gut Lipidome; Skin Lipidome; Blood Lipidome
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): • Probiotic fomula per capsule:
  2 Billion CFUs HU36 - 30 mg HU58 - 20 mg Bacillus clausii -25 mg Bacillus coagulans 10B - 35 mg Prepro - 22 mg. The prebiotic that is to be used in the proprietary blend is a vegetable grade cellulose.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Rice flour only
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — • Probiotic fomula per capsule:
  * 2 Billion CFUs
  * HU36 - 30 mg
  * HU58 - 20 mg
  * Bacillus clausii -25 mg
  * Bacillus coagulans 10B - 35 mg
  * Prepro - 22 mg. The prebiotic that is to be used in the proprietary blend is a vegetable grade cellulose.
  Arms: Probiotic
Other: Placebo — Rice flour only
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure oil production of the face, facial properties, and gut bacteria in people being given oral probiotics. Probiotic supplements contain active cultures of bacteria that are thought to be beneficial to human health.The investigators want to find out if probiotics taken by mouth alter the bacteria in subject's gut and subject's skin oil production compared to a placebo. This is a single blind study and subject may receive a probiotic or a placebo for the first half of the study and a placebo or a probiotic for the second half of the study. Subject will not know what was given to participants.

DETAILED DESCRIPTION:
Antibiotics are widely used within dermatology for the treatment of chronic skin conditions such as acne, rosacea, and atopic dermatitis. Previous studies have shown that oral probiotics may be beneficial for skin disesaes such as atopic dermatitis and acne, but a mechanism for how the gut communicates to the skin remains elusive.

The balance between short chain fatty acids and long chain fatty acids has been proposed as one factor in how bacteria in the gut are able to communicate with the rest of the body. Studies in Dr. Sivamani's lab have shown that subjects with acne have a reduced level of short chain fatty acids in their blood when compared to age-matched control (unpublished).

The aim of this study is to understand how oral probiotics may alter the gut microbiome and if they can augment the short chain fatty acids in the blood lipidome. Ultimately, the investigator's goal is to find suitable alternatives for the use of antibiotics in the treatment of chronic skin conditions so that the amount of antibiotics that are in use can be reduced.

ELIGIBILITY:
Inclusion Criteria

• 18 years of age or older

Exclusion criteria

* Those on oral antibiotics within a month of initiating the study.
* Subjects must have no history of diabetes, known cardiovascular disease, known immunocompromised condition, malignancy, kidney disease, or chronic steroid use.
* Subjects must have no history or diagnosis of gastrointestinal inflammatory diseases.
* Those with BMI higher than 30 kg/m²
* Those on topical medications to the face such as retinoids or antibiotics who are not willing or medical unable (in the judgement of the investigator) to discontinue use for two weeks prior to the study and for the duration of study participation.
* Those that have undergone a change in hormonally based therapies, such as but not limited to oral contraceptive pills or progesterone based pills within the last two months. Progesterone releasing IUDs are considered hormone releasing therapy.
* Use of medications that alter blood lipids, such as statins and anti-hyperlipidemic medications
* Current tobacco smokers, OR those that have smoked tobacco over the past year, OR a 5 year-pack year history of smoking tobacco
* Pregnant women
* Prisoners
* Adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Blood Lipidome Changes | 8 weeks +/- 1 week
  The primary objective is to assess if probiotics rich in the production of short chain fatty acids can shift the blood lipidome to have a higher level of short chain fatty acids

SECONDARY OUTCOMES:
Gut Microbiome Changes | 8 weeks +/- 1 week
  Specifically the presence of short chain fatty acid producing bacteria
Sebum Production | 8 weeks +/- 1 week
  Sebum production will be measured via Sebumeter device that will calculate sebum in micrograms/centimeter^2
Hydration | 8 weeks +/- 1 week
  Hydration will be measured via Moisturemeter device that will measure hydration in arbitrary units (AU)

CONTACTS AND LOCATIONS:
Overall Officials: Raja K. Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided